CLINICAL TRIAL: NCT03023111
Title: Miltefosine and GM-CSF in Cutaneous Leishmaniasis: a Randomized and Controlled Trial
Brief Title: Miltefosine and GM-CSF in Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, MD, PhD, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mil GM CL-2017
Record Dates: First submitted 2016-12-27; First posted 2017-01-18 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous leishmaniasis; miltefosine; cytokines; treatment
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate; miltefosine; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sbv (Active Comparator): Meglumine antimoniate (Glucantime):
  Dosage: 20 mg / kg / day, intravenously, during 20 days.
  Interventions: Drug: Sbv
- Miltefosine plus placebo (Experimental): Miltefosine (28 days / 2.5mg / Kg / day at a maximum dose of 150mg / day orally) + Topical placebo (gel cream, 2 times a day for 28 days)
  Interventions: Drug: Miltefosine plus placebo
- Miltefosine plus GM-CSF (Experimental): Miltefosine (28 days / 2.5mg / kg / day at a maximum dose of 150mg / day orally) + Topical GM-CSF (0.01% gel cream, 2 times a day for 28 days)
  Interventions: Drug: Miltefosine plus GM-CSF

INTERVENTIONS:
Drug: Sbv — Standard treatment for CL, parenteral drug used during 20 days.
  Other Names: Glucantime
  Arms: Sbv
Drug: Miltefosine plus placebo — Oral treatment for CL, capsules with 50mg used 3 times a day, during 28 days. Placebo gel cream will be used topically.
  Other Names: Impavido plus placebo
  Arms: Miltefosine plus placebo
Drug: Miltefosine plus GM-CSF — Oral treatment for CL, capsules with 50mg used 3 times a day, during 28 days. GM-CSF gel cream will be used topically.
  Other Names: Impavido plus GM-CSF
  Arms: Miltefosine plus GM-CSF

SUMMARY:
Cutaneous leishmaniasis (CL) standard treatment is done with parenteral pentavalent antimony (Sbv) at the dose of 15-20mg / kg per day for 20 days. However, therapeutic failure has been described in up to 50% of patients, and the long period of 60 to 90 days required for healing of the ulcerated lesion indicate the need for alternative drugs. Currently the alternatives include other parenteral drugs such as pentamidine and amphotericin B, whose use is limited either by toxicity or because, as with Sbv, the parenteral route hinders adherence and regularity of treatment in the rural area. Recent studies by our group indicate that oral miltefosine is the most effective drug for the treatment of patients with CL caused by L. (V.) guyanensis and L. (V.) braziliensis in Brazil, with a cure rate of 71.4% and 75% respectively. CL pathogenesis is associated with intense inflammatory infiltrate and tissue damage. Previous trials associating GM-CSF to Sbv improved the cure rate of CL caused by L. (V.) braziliensis. The objective of this trial is to evaluate the therapeutic response to the use of miltefosine associated to GM-CSF in the treatment of CL caused by L. (V.) braziliensis in an endemic region in Bahia and Ceará, and by L. (V.) guyanensis in the Amazon region.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated ulcerative cutaneous leishmaniasis, with laboratory diagnosis obtained through at least one of the following tests: direct examination of the lesion, positive culture or PCR for Leishmania.
2. Age: 18 to 65 years;
3. Sex: male and female patients;
4. Presence of at least 1 ulcerated lesion at any location;
5. Presence of a maximum of 3 ulcerated lesions;
6. Diameter of lesions varying between 1 and 5 cm;
7. Clinical evolution of the disease of not less than 1 month and not more than 3 months.

Exclusion Criteria:

1. Evidence of severe underlying disease (cardiac, renal, hepatic, pulmonary) or malignant disease;
2. Patients with immunodeficiency or HIV carriers;
3. Serious protein and / or caloric malnutrition;
4. Active and uncontrolled infectious-contagious disease such as tuberculosis, leprosy, systemic fungal disease (histoplasmosis, paracoccidioidomycosis) or any other similar condition;
5. Women who are pregnant or breastfeeding;
6. Allergy to Sbv or miltefosine;
7. Previous treatment for leishmaniasis;
8. Lack of capacity or willingness to provide informed consent (patient and / or parent / legal representative); Absence of availability for the visits or to comply with the study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Final cure rate or complete cicatrization of the ulcer | 6 months after the end of treatment
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients. Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.

SECONDARY OUTCOMES:
Initial cure rate or initial cicatrization of the ulcer | 2 months after the end of treatment
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients. Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.
Healing time | Up to 2 months after the end of treatment
  Time (in days) to achieve complete cicatrization will be recorded.
Clinical and laboratory adverse events | During treatment and through study completion, an average of 1 year
  Clinical and laboratory adverse events will be recorded and graded according to the Common Terminology Criteria for Adverse Event (CTCAE) of the National Cancer Institute

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RL Machado, MD, PhD, Principal Investigator — Federal University of Bahia; Edgar M Carvalho, MD, PhD, Study Director — Instituto Fernandes Figueira; Manoel Barral Neto, MD, PhD, Study Chair — Instituto Fernandes Figueira; Gerson Penna, MD, PhD, Study Chair — Instituto Fernandes Figueira
Locations (2):
- Brazil (2):
  - Fundação de Medicina Tropical do Amazonas, Manaus, Amazonas
  - Corte de Pedra Health Post, Presidente Tancredo Neves, Estado de Bahia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendes L, Guerra JO, Costa B, Silva ASD, Guerra MDGB, Ortiz J, Doria SS, Silva GVD, de Jesus DV, Barral-Netto M, Penna G, Carvalho EM, Machado PRL. Association of miltefosine with granulocyte and macrophage colony-stimulating factor (GM-CSF) in the treatment of cutaneous leishmaniasis in the Amazon region: A randomized and controlled trial. Int J Infect Dis. 2021 Feb;103:358-363. doi: 10.1016/j.ijid.2020.11.183. Epub 2020 Nov 27. PMID 33253864
- [Derived] Machado PRL, Prates FVO, Boaventura V, Lago T, Guimaraes LH, Schriefer A, Corte TWF, Penna G, Barral A, Barral-Netto M, Carvalho EM. A Double-blind, Randomized Trial to Evaluate Miltefosine and Topical Granulocyte Macrophage Colony-stimulating Factor in the Treatment of Cutaneous Leishmaniasis Caused by Leishmania braziliensis in Brazil. Clin Infect Dis. 2021 Oct 5;73(7):e2465-e2469. doi: 10.1093/cid/ciaa1337. PMID 32894278